CLINICAL TRIAL: NCT03865732
Title: A Double-blind, Randomized, Placebo-controlled Trial of Adjunctive Ganaxolone Treatment in Female Children With Protocadherin 19 (PCDH19)-Related Epilepsy Followed by Long-term Open-label Treatment.
Brief Title: Study of Adjunctive Ganaxolone Treatment in Female Children With Protocadherin 19 (PCDH19)-Related Epilepsy (Violet Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-PCDH19-3002; 2018-004496-12 (EudraCT Number)
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Results first posted 2022-09-08 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: PCDH19-Related Epilepsy
Keywords: refractory seizures; epilepsy in children; seizure disorder
MeSH Terms: conditions — Seizures; Epilepsy | interventions — ganaxolone

STUDY DESIGN:
Intervention Model Description: The double-blind phase will randomize subjects to adjunctive ganaxolone or placebo at a 1:1 ratio to standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo suspension 3x's /day for 17 weeks
  Interventions: Drug: Placebo
- Ganaxolone (Experimental): ganaxolone suspension (50 mg/ml) 3x's /day for 17 weeks
  Interventions: Drug: Ganaxolone

INTERVENTIONS:
Drug: Ganaxolone — active drug
  Arms: Ganaxolone
Drug: Placebo — inactive
  Other Names: Placebo (for ganaxolone)
  Arms: Placebo

SUMMARY:
A clinical study to evaluate the efficacy, safety, and tolerability of adjunctive ganaxolone therapy compared to placebo for the treatment of seizures in female children and young adults with genetically confirmed PCDH19 gene mutation.

DETAILED DESCRIPTION:
The Violet Study is a global, double-blind, placebo-controlled, Phase 2 clinical trial that plans to enroll approximately 25 female patients between the ages of 1 and 17 with a confirmed disease-related PCDH19 gene variant. Patients will undergo a baseline period before being randomized to receive, in addition to their existing anti-seizure treatment, either ganaxolone or placebo for 17 weeks. Following the treatment period, all patients that meet certain eligibility requirements will have the opportunity to receive ganaxolone in the open label phase of the study. The study's primary efficacy endpoint is percent reduction in seizures. Secondary outcome measures will include non-seizure-related endpoints to capture certain behavioral and sleep disturbances that have been seen in previous clinical studies with ganaxolone.

ELIGIBILITY:
Inclusion Criteria:

* Molecular confirmation of a pathogenic or likely pathogenic PCDH19 variant
* Failure to control seizures despite 2 or more anti-seizure medications
* 12 seizures over a 12-week period of primary seizure types prior to screening
* On a stable regimen of concomitant AEDs, Ketogenic diets, and modified Atkins diet should be unchanged for 3 months prior to screening)

Exclusion Criteria:

* Previous exposure to ganaxolone
* > 8 consecutive weeks of seizure freedom during the 12 weeks prior to screening
* Concurrent use of strong inducers or inhibitors of CYP3A4/5/7 is not permitted
* Use of tetrahydrocannabinol (THC) or non-approved cannabidiol (CBD) is prohibited during the double-blind phase
* Exposure to any other investigational drug within 30 days or fewer than 5 half-lives prior to screening

Ages: 1 Year to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2022-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Gasior, M.D., Ph.D, Study Director — Marinus Pharmaceuticals, Inc.; Paula Bokesk, M.D., FAAP, Study Director — Marinus Pharmaceuticals, Inc.
Locations (12):
- United States (6):
  - Marinus Research Site, Little Rock, Arkansas
  - Marinus Research Site, Los Angeles, California
  - Marinus Research Site, San Francisco, California
  - Marinus Research Site, Durham, North Carolina
  - Marinus Research Site, York, Pennsylvania
  - Marinus Research Site, Salt Lake City, Utah
- Marinus Research Site, Budapest, Hungary
- Italy (2):
  - Marinus Research Site, Florence
  - Marinus Research Site, Rome
- Netherlands (2):
  - Marinus Research Site, Heeze
  - Marinus Research Site, Zwolle
- Marinus Research Site, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sullivan J, Gunning B, Zafar M, Guerrini R, Gecz J, Kolc KL, Zhao Y, Gasior M, Aimetti AA, Samanta D. Phase 2, placebo-controlled clinical study of oral ganaxolone in PCDH19-clustering epilepsy. Epilepsy Res. 2023 Mar;191:107112. doi: 10.1016/j.eplepsyres.2023.107112. Epub 2023 Feb 22. PMID 36870093

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo suspension 3x's/day for 17 weeks
Period: Overall Study
Arm/Group | Placebo | Ganaxolone
Started | 11 | 10
Completed | 11 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Placebo: placebo suspension 3x's /day for 17 weeks
  Placebo: non-active drug
- Total: Total of all reporting groups
Arm/Group | Placebo | Ganaxolone | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (3.93) | 6.7 (3.40) | 7.1 (3.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 7 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 2 | 2 | 4
  Hungary | 1 | 0 | 1
  United States | 6 | 6 | 12
  Poland | 0 | 2 | 2
  Italy | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Summary of 28-day Seizure Frequency Through 17 Week Post-Baseline Phase (Median Percent Change)
Description: Summary of 28-Day Seizure Frequency for Seizure Types through 17 week Post-Baseline Phase (Median Percent Change)
Time Frame: End of the double-blind 17 week treatment period
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: Median % Change in Number of Seizures
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 11 | 10
Median % Change in Number of Seizures | -23.97 [-88.24 to 4.89] | -61.52 [-95.85 to -33.40]

2. Secondary Outcome: Summary of 28-day Seizure Frequency for Subjects in the Biomarker-positive Stratum (Median Percent Change)
Description: Summary of 28-day Seizure Frequency for Seizure Types for Subjects in the Biomarker-positive Stratum through 17 weeks (Median Percent Change)
Time Frame: [Time Frame: End of the double-blind 17 week treatment period]
Population: ITT Population specific to subjects in the Biomarker-positive Stratum
Measure: Median (Inter-Quartile Range); unit: Median % Change in Number of Seizures
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 7 | 6
Median % Change in Number of Seizures | -18.71 [-85.74 to 70.73] | -35.90 [-86.48 to -24.32]

3. Secondary Outcome: 50% Primary Seizure Reduction
Description: Percent of subjects experiencing a greater than or equal to 50% reduction in 28-day primary seizure frequency relative to the 12-week baseline
Time Frame: End of the double-blind 17 week treatment period
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 11 | 10
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: Screening through Week 17
Arm/Group | Placebo | Ganaxolone
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/11 | 1/10
Other Adverse Events (participants affected / at risk) | 11/11 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Ganaxolone (N=10)
Psychogenic Seizure (Psychiatric disorders) | 0 (0) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 1 (3) | 0 (0)
Seizure (Nervous system disorders) | 3 (4) | 0 (0)
Seizure Cluster (Nervous system disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Ganaxolone (N=10)
Aggression (Psychiatric disorders) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Behavior Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Psychogenic Seizure (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1)
Disinhibition (Psychiatric disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 4 (4)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (5) | 0 (0)
Seizure Cluster (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2)
Gait Disturbance (General disorders) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2)
Protein Urine Present (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT03865732/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT03865732/SAP_003.pdf